CLINICAL TRIAL: NCT02106598
Title: Targeted Silica Nanoparticles for Real-Time Image-Guided Intraoperative Mapping of Nodal Metastases
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-249
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Melanoma
Keywords: Sentinel Lymph Node Mapping; Intraoperative Sentinel; Head and Neck Melanoma; Targeted Silica Nanoparticles; cRGDY-PEG-Cy5.5-C dots; 13-249

ARMS (1):
- Phase 2 - Head and Neck Cancer (Experimental): Patients with early oral cavity squamous cell carcinoma, and prior to standard of care wide local resection of the primary tumor and elective neck dissection, will receive a locally-administered, peritumoral injection of fluorescent cRGDY-PEG-Cy5.5-C dots (0.25 - 1 ml) around the primary lesion while under standard-of-care anesthesia for identification of optically-avid SLNs and to assess for metastatic disease. After completion of the neck dissection, nodal specimens will be examined ex vivo for fluorescence signal. Any fluorescent and non-fluorescent nodes will be compared to determine the true positive and false positive rates for cancer detection in this pilot study. No change in standard of care surgical practice will occur.
  Interventions: Drug: fluorescent cRGDY-PEG-Cy5.5-C dots

INTERVENTIONS:
Drug: fluorescent cRGDY-PEG-Cy5.5-C dots

SUMMARY:
Current imaging devices usually detect cancer prior to surgery. However, these devices cannot be used during the surgical procedure to visualize lymph nodes with cancer (called "sentinel lymph nodes"). This is a Phase II study, containing a total of 67 patients with head and neck cancer. The purpose of this study is to test if imaging, with cRGDY-PEG-Cy5.5-C dots is useful for evaluating your type of cancer. This is currently not approved by the FDA. The researchers want to see if cRGDY-PEG-Cy5.5-C dots, can improve upon the usual scans. As a part of your standard of care, you will initially undergo imaging of your lymph nodes prior to your surgery. Prior to your surgery, you will be injected with a radioactive dye around the tumor site, and images will be acquired about 2 hours later using a device to image the location of the dye. We have tested, for the first time in humans, a new, experimental dye-labeled particle (dots), cRGDY-PEG-Cy5.5-C dots for lymph node mapping. This particle, the size of a small protein, will be injected around sites of your tumor before or during your surgery to identify diseased nodes using a hand-held camera system. The dye-labeled particle can be viewed in tissues that may contain tumor. The particles will not treat your cancer and any images or information found during this study will not be used for your treatment. The information collected may be used to guide the design of future studies to detect and/or treat tumors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed diagnosis of melanoma at MSKCC
* Have one of the following disease histories:
* Newly-diagnosed or recurrent (local, regional, metastatic) malignant melanoma, oral cavity squamous cell carcinoma, and squamous cell carcinoma of the skin patients in whom SLN mapping is indicated

  * Residual clinically or radiographically evident tumor, including primary cutaneous and mucosal melanomas
  * Prior radiation therapy, chemotherapy, or surgery in patients requiring flap reconstruction in the head and neck region.
  * Newly diagnosed patients with previous excisional biopsy.
* At the discretion of the physician or surgeon, normal baseline cardiac function based upon pre-operative evaluation
* At the discretion of the operating surgeon, ANC>1000/mcl and platelets>100,000/mcl.
* At the discretion of the physician or surgeon, bilirubin level of < 2.0 mg/dl in the absence of a history of Gilbert's disease (or pattern consistent with Gilbert's).
* For melanoma patients, if patients have a history of malignancy other than melanoma, and other skin cancers in the past five years, their inclusion is up to the discretion of the physician.
* All patients of childbearing and child-creating age must be using an acceptable form of birth control
* Women who are pre-menopausal must have a negative serum pregnancy test

Exclusion Criteria:

* Known pregnancy or breast-feeding.
* Medical illness unrelated to the tumor which in the opinion of the attending physician and principal investigator will preclude administration of the agent. This includes patients with uncontrolled infection, chronic renal insufficiency, myocardial infarction within the past 6 months, unstable angina, cardiac arrhythmias other than chronic atrial fibrillation and chronic active or persistent hepatitis, or New York Heart Association Classification III or IV heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
feasibility of conducting pre-operative SLN mapping | 1 year
  using real-time optical detection procedures and intradermal single- or double-dose injection/s of non-radioactive cRGDY-PEG-Cy5.5-C dots about the primary tumor site. Feasibility will be determined on the basis of achieving adequate image contrast for detection, as defined by signal-to-background ratios, and whether optical signal distinguishes diseased SLNs from non-diseased ones

CONTACTS AND LOCATIONS:
Overall Officials: Hilda Stambuk, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York

REFERENCES:
- [Derived] Zanoni DK, Stambuk HE, Madajewski B, Montero PH, Matsuura D, Busam KJ, Ma K, Turker MZ, Sequeira S, Gonen M, Zanzonico P, Wiesner U, Bradbury MS, Patel SG. Use of Ultrasmall Core-Shell Fluorescent Silica Nanoparticles for Image-Guided Sentinel Lymph Node Biopsy in Head and Neck Melanoma: A Nonrandomized Clinical Trial. JAMA Netw Open. 2021 Mar 1;4(3):e211936. doi: 10.1001/jamanetworkopen.2021.1936. PMID 33734415
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/